CLINICAL TRIAL: NCT04549857
Title: The Effects of Aromatherapy on Pain, Sleep Quality, and Psychological Distress in Patients With Rheumatoid Arthritis.
Brief Title: Effects of Aromatherapy on Pain, Sleep Quality, and Psychological Distress in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TYGH108056
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
Keywords: aromatherapy; rheumatoid arthritis; pain; sleep quality; psychological distress
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain; Sleep Initiation and Maintenance Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Experimental): The experimental group used the base oil (sweet almond oil) to add Atlantic cedar, sweet marjoram and sweet orange essential oils. The essential oils were blended into 5% massage oil at a ratio of 3:1:1.
  Interventions: Behavioral: aromatherapy
- Placebo group (Placebo Comparator): The placebo group only used base oil (sweet almond oil).
  Interventions: Behavioral: aromatherapy
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: aromatherapy — The intervention measures were taught by the researchers to perform self-massage on both wrists and finger joints in the experimental group and the comfort group, using 5ml each time (2.5ml each for one hand), 10 minutes each time (5 minutes for each hand), three times a week, It lasts for three weeks. The massage steps refer to dōTERRA's Aroma Touch Hand Technique. Before self-massage is performed, a professional must first ensure that the execution process is correct and the professional will use the phone to follow up weekly.
  1. The experimental group used the base oil (sweet almond oil) to add Atlantic cedar, sweet marjoram and sweet orange essential oils. The essential oils were blended into 5% massage oil at a ratio of 3:1:1.
  2. The placebo group only used base oil (sweet almond oil).
  3. The control group did not provide any interventional measures and only received conventional treatment.
  Arms: Placebo group; intervention group

SUMMARY:
This study aims to explore the effects of aromatherapy on pain, sleep quality, and psychological distress in patients with rheumatoid arthritis. The following hypotheses are tested: The experimental group received aromatherapy will report significant improvement on pain, sleep quality, and psychological distress.The comfort group shows no significant differences.

DETAILED DESCRIPTION:
The purpose of the research was to explore the effects of aromatherapy on pain, sleep quality, and psychological distress in patients with rheumatoid arthritis. The subjects of the study adopted the intentional sampling method, and the place of collection was patients with rheumatoid arthritis in the outpatient department of the rheumatology and immunology department of the hospital. The study was conducted with a randomized controlled trial design. It is estimated that 159 patients with rheumatoid arthritis will be admitted, and the participants will be randomly allocated into the experimental group, the comfort group and the control group with 53 participants. The experimental group received base oil and essential oil massage, the comfort group only received base oil massage for 10 minutes each time, three times a week for three weeks, and the control group did not receive any intervention measures. Repeated measurements were used to collect data using structured questionnaires. Pain was measured by the Numerical Rating Scale, and sleep quality was measured by the Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale. Scale) measurement and psychological distress were measured by the Hospital Anxiety and Depression Scale. Data were collected at four time points before the intervention, the first week, the second week, and the third week after the intervention. The data obtained are processed and analyzed using SPSS version 22.00 computer software. Statistical analysis methods include independent sample single-factor variance analysis to compare the differences in basic data and pain levels between the experimental group, the comfort group and the control group; repeated measurement of single-factor variation Analyze the comparison of intra-group differences among the three groups at four time points; finally, compare the effects of the three groups on pain and sleep quality after aromatherapy interventions using the generalized estimation equation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by a doctor as rheumatoid arthritis.
* Over 20 years old.
* No history of allergy to essential oils in the past.
* A person with clear consciousness and able to communicate in Mandarin or Taiwanese.
* Those who are willing to participate in this research after the explanation.
* The main part of the pain in the past month is the joints of the hand.
* Have equipment that can watch movies.

Exclusion Criteria:

* There is a history of wounds or surgery around the wrist or finger joints.
* Those who are contraindicated in aromatherapy and those with high risk such as asthma, epilepsy, and pregnant.
* Receive physical therapy or complementary therapy during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Numerical Rating Scale scores | 1 week, 2 weeks and 3 weeks
  Change from baseline Pain Numerical Rating Scale scores at 1 week, 2 weeks and 3 weeks. The total score range is 0-10; a higher score indicates more pain
Changes in Pittsburgh Sleep Quality Index scores | 1 week, 2 weeks and 3 weeks
  Change from baseline Pittsburgh Sleep Quality Index scores at 1 week, 2 weeks and 3 weeks. The total score range is 0-21; a higher score indicates poor sleep

SECONDARY OUTCOMES:
Changes in Hospital Anxiety and Depression Scale scores | 1 week, 2 weeks and 3 weeks
  Change from baseline Hospital Anxiety and Depression Scale scores with two subscales at 1 week, 2 weeks and 3 weeks. Each subscale score range is 0-21; a higher score indicates higher anxiety and depression.
Changes in Epworth Sleepiness Scale scores | 1 week, 2 weeks and 3 weeks
  Change from baseline Epworth Sleepiness Scale scores at 1 week, 2 weeks and 3 weeks. The total score range is 0-24; a higher score indicates more sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No